CLINICAL TRIAL: NCT04789798
Title: The Efficiency of Telemedicine to Optimize Metabolic Control in Patients With Diabetes in Turkey: Preliminary Results From The Randomised Controlled Telediab Trial
Brief Title: The Efficiency of Telemedicine to Optimize Metabolic Control in Patients With Diabetes in Turkey
Acronym: TELEDIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Turker, MD, PhD; Academician; Principle Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012/1461-1217
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Telemedicine; Telehealth
Keywords: Telemedicine; Telehealth; Virtual care; Diabetes; Virtual visits
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TeleDiab (Telemedicine) (Experimental): TeleDiab program components consist of:
  1. Electronic transmission of capillary blood glucose measurement results
  2. Electronic transmission of blood pressure measurements
  3. Synchronized video-conferencing, secure messaging
  4. Access to clinical data from patient files when necessary
  5. Reminding of routine follow-up tests and examinations
  6. Providing web-based educational materials to patients.
  Interventions: Device: TeleDiab (Telemedicine)
- Usual Care (Active Comparator): usual diabetes care, as provided by primary care providers in the hospital
  Interventions: Other: Usual care

INTERVENTIONS:
Device: TeleDiab (Telemedicine) — TeleDiab program components consist of:
  1. Electronic transmission of capillary blood glucose measurement results
  2. Electronic transmission of blood pressure measurements
  3. Synchronized video-conferencing, secure messaging
  4. Access to clinical data from patient files when necessary
  5. Reminding of routine follow-up tests and examinations
  6. Providing web-based educational materials to patients.
  Arms: TeleDiab (Telemedicine)
Other: Usual care — Usual diabetes care, as provided by primary care providers
  Arms: Usual Care

SUMMARY:
The direct and indirect costs of treating diabetes are high. 10-15% of the health budgets of many countries are spent on diabetes treatment. Most of these expenses are due to the treatment and follow-up costs of complications seen in patients who are not well monitored and whose metabolic control is not achieved. the rapid increase in diabetes causes polyclinic and hospital services to become more intense. Despite the increasing number of patients, both performance and due to non-physician occupational groups' insufficiency (Diabetes Dietician, Diabetes Nurse), patients can only be given an appointment once a year, and patients cannot be allocated sufficient time during the appointment. Since these problems are valid worldwide, Telemedicine programs are designed to provide easy, cheap, and practical follow-up and treatment of many chronic diseases in various states of the USA and many developed European countries.

DETAILED DESCRIPTION:
The project is designed as a randomized controlled trial with approximately 100 subjects receiving a telemedicine intervention and approximately 100 receiving usual care. Eligibility requires having diabetes and being a Medicare beneficiary.

This program, called "TeleDiab" for the first time in our country, was designed in cooperation with the Istanbul University Rectorate and the local telecommunication company Turkcell. Its implementation was carried out as a pilot project in the Department of Endocrinology and Metabolic Diseases of Istanbul Medical Faculty in the follow-up and treatment of diabetic patients. Subjects are randomized to receive telemedicine case management or usual care for diabetes.

This project, it is aimed to evaluate the "TeleDiab" program developed for use in diabetic patients in terms of applicability, practicality, effectiveness, and cost-effectiveness. In this way, it was aimed to compare the electronically followed patient group with a similar patient group routinely followed in terms of glycemic control, treatment compliance, complications, and comorbid diseases 6 months and 1 year later.

The intervention utilizes a home telemedicine unit (HTU). The HTU is a specially designed, web-enabled device with a data port connected to a home glucometer and home blood pressure cuff whereby measurements obtained with these devices can be directly uploaded to a computer database. A diabetes nurse and a practitioner case manager interact regularly with intervention participants through videoconference via the HTU.

ELIGIBILITY:
Inclusion Criteria:

for TeleDiab group:

* Have known Type 1 diabetes for at least 3 months or Type 2 diabetes using basal-bolus insulin
* Being between the ages of 18-65
* Istanbul University Istanbul Medical Faculty Internal Diseases Department, Endocrinology and Being registered and being monitored in the Metabolic Diseases BD, Diabetes Outpatient Clinic
* To be able to measure blood glucose from the fingertip (couplings) at home
* To be able to measure blood pressure at home
* To be able to use computers and smartphones
* Instead of electronic directives and recommendations of the physician or diabetes nurse be able to bring
* Agree to participate in the study.

for the control group:

* Have known Type 1 diabetes for at least 3 months or Type 2 diabetes using basal-bolus insulin
* Being between the ages of 18-65
* Istanbul University Istanbul Medical Faculty Internal Diseases Department, Endocrinology and Being registered and being monitored in the Metabolic Diseases BD, Diabetes Outpatient Clinic
* Inability to use computer and smartphone
* Failure to follow the electronic directives and recommendations of the physician or diabetes nurse

Exclusion Criteria:

* <18 and> 65years old
* Presence of Type 1 diabetes for less than 3 months or Type 2 diabetes not using insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2015-10-19 (Actual); Study Completion 2015-10-19 (Actual)

PRIMARY OUTCOMES:
Capillary glucose levels changes | Change in baseline capillary glucose levels (mg/dl) at 24th month
Home blood glucose measurement frequency | Change in baseline home blood glucose measurement frequency at 24th month
A1c measurement | Change in baseline A1c (%) measurement frequency at 24th month
Weight | Change in baseline weight (kg) measurement frequency at 24th month
BMI | Change in baseline BMI (kg/m2) measurement frequency at 24th month

SECONDARY OUTCOMES:
Number of patients developing new diabetes complications within 24 months | Change from baseline to 24 months
  retinopathy, peripheral neuropathy, autonomic neuropathy, nephropathy
Number of patients who developed new comorbidities in 24 months | Change from baseline to 24 months
  hyperlipidemia, hypertension, coronary artery disease, stroke, peripheral artery disease, general obesity, central obesity, clinical or subclinical hypo or hyperthyroidism, autoimmune trioiditis, celiac disease; gluten enteropathy, other
The number of patients who added insulin to their oral antidiabetic medication or switched to oral antidiabetic medication by discontinuing insulin | Change from baseline to 24 months

OTHER OUTCOMES:
Serum ALT levels | Change from baseline to 24 months
Serum TSH levels | Change from baseline to 24 months
Serum sT4 levels | Change from baseline to 24 months
Serum LDL levels | Change from baseline to 24 months
Serum HDL levels | Change from baseline to 24 months
Serum triglyceride levels | Change from baseline to 24 months
Serum BUN levels | Change from baseline to 24 months
Serum creatinine levels | Change from baseline to 24 months
Serum hemoglobine levels | Change from baseline to 24 months
eGFR levels | Change from baseline to 24 months
Urine microalbuminurea | Change from baseline to 24 months

REFERENCES:
- [Background] Shea S, Weinstock RS, Teresi JA, Palmas W, Starren J, Cimino JJ, Lai AM, Field L, Morin PC, Goland R, Izquierdo RE, Ebner S, Silver S, Petkova E, Kong J, Eimicke JP; IDEATel Consortium. A randomized trial comparing telemedicine case management with usual care in older, ethnically diverse, medically underserved patients with diabetes mellitus: 5 year results of the IDEATel study. J Am Med Inform Assoc. 2009 Jul-Aug;16(4):446-56. doi: 10.1197/jamia.M3157. Epub 2009 Apr 23. PMID 19390093